CLINICAL TRIAL: NCT02207855
Title: Chloroprocaine for Continuous Epidural Analgesia in Neonates and Infants
Status: Completed | Type: Observational
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB14-00231
Record Dates: First submitted 2014-08-01; First posted 2014-08-04 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Anesthesia
MeSH Terms: interventions — chloroprocaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chloroprocaine: Neonates and infants who have received chloroprocaine for epidural anesthesia.
  Interventions: Drug: Chloroprocaine

INTERVENTIONS:
Drug: Chloroprocaine

SUMMARY:
This a study to retrospectively review our experience with the use of chloroprocaine for postoperative epidural infusions in neonates and infants. Pain scores and the need for intravenous analgesic agents will be recorded from the records to demonstrate the efficacy of the technique.

ELIGIBILITY:
Inclusion Criteria:

* Neonates and infants who have received chloroprocaine for epidural anesthesia.

Exclusion Criteria:

* None

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates and infants who have received chloroprocaine for epidural anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Pain score | Every 6 hours for 72 hours

SECONDARY OUTCOMES:
Pain medicine consumption | Every 6 hours for 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tobias, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States